CLINICAL TRIAL: NCT06049901
Title: Clinical Study Evaluating the Efficacy and Safety of Nitazoxanide in Patients With Metastatic Colorectal Cancer
Brief Title: Nitazoxanide in Patients With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reham Ameen El-Ghoneimy, Assistant Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nitazoxanide in mCRC
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Nitazoxanide
MeSH Terms: conditions — Colorectal Neoplasms | interventions — nitazoxanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will include 30 patients who will be scheduled to receive 6 cycles of 5-Fluorouracil and Oxaliplatin- based regimens every 2 weeks for 3 months.
- Nitazoxanide Group (Active Comparator): This group will include 30 patients who will be scheduled to receive 6 cycles of 5-Fluorouracil and Oxaliplatin- based regimens every 2 weeks plus nitazoxanide (500 mg orally twice daily) for 3 months.
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — Nitazoxanide is considered a broad-spectrum anti-microbial drug with a potent activity against various helminths, anaerobic bacteria and viruses.
  Other Names: Nanazoxid
  Arms: Nitazoxanide Group

SUMMARY:
The aim of this study is to evaluate the potential efficacy and safety of nitazoxanide in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Globally, colorectal cancer (CRC) is a major malignant tumor of the gastrointestinal tract which originates from epithelial cells of the colon and rectum. The efficacy of current cancer therapies is still limited by severe adverse effects on normal tissues and chemoresistance development. Therefore, recent efforts have been focused on the repurposing of existing drugs with good safety profiles for cancer treatment.

Nitazoxanide (NTZ) is considered a broad-spectrum anti-microbial drug with a potent activity against various helminths, anaerobic bacteria and viruses. NTZ inhibited the proliferation of CRC cell lines at or below concentrations that normally exhibit anti-parasitic activity.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage IV (metastatic) CRC. Staging will be performed according to the American Joint Committee on Cancer (AJCC) 8th edition and will be documented by all investigating parameters of metastatic CRC
2. Male or female patients with age range from 18-65 years old
3. Women of childbearing age will be required to be on acceptable forms of contraception
4. No contraindication to chemotherapy (absence of myelosuppression)
5. Performance status < 2 according to the Eastern Cooperative Oncology Group (ECOG) score
6. Adequate liver function (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < grade 2) according to the National Cancer Institute-Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v 5.0)
7. Adequate renal function (estimated creatinine clearance (eCrCl), serum creatinine (SCr) < grade 2) according to NCI-CTCAE, v 5.0
8. Adequate hematological parameters (hemoglobin, erythrocytes, platelets, leukocytes and absolute neutrophil count (ANC) < grade 2 according to NCI-CTCAE, v 5.0

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients who have known allergy to nitazoxanide or its metabolites
3. Patients with concurrent active cancer originating from a primary site other than the colon or rectum
4. Patients who are receiving highly plasma protein-bound drugs or drugs with extensive hepatic metabolism such as; coumarin anti-coagulants, oral hypoglycemic drugs and anti-epileptic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Investigating the possible efficacy of nitazoxanide through evaluation of its impact on overall response rate (ORR) and disease control rate (DCR). | 3 months
  Abdominal, pelvic and chest CT scanning will be performed at baseline and after 3 months. ORR and DCR will be evaluated and categorized according to the RECIST 1.1 criteria. ORR includes patients with both complete response and partial response. DCR includes patients with complete response, partial response and stable disease. Both ORR and DCR will be determined as number and percentage.
Evaluating the change in the serum level of Reduced glutathione (GSH) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Superoxide dismutase (SOD) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Nuclear factor-kappa B (NF-kB) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Protein disulfide isomerase (PDI) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.

SECONDARY OUTCOMES:
Evaluating the one-year overall survival (1-year OS) | 12 months
  OS is defined as the time from randomization to death from any cause is OS. One-year OS will be determined as mean and median in months.
Evaluating the progression free survival (PFS) | 12 months
  PFS is defined as the time from randomization to investigator- assessed tumor progression. PFS will be determined as mean and median in months.
Evaluating the safety and tolerability of nitazoxanide through investigating Liver function test (ALT (U/mL) and AST (U/mL)). | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.
Evaluating the safety and tolerability of nitazoxanide through investigating Renal function test (SCr (mg/dL), BUN (mg/dL) and eCrCl (mL/min)). | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.
Evaluating the safety and tolerability of nitazoxanide through investigating Hematological parameters (hemoglobin (mg/dL), erythrocytes (cells/μL), leukocytes (cells/μL), platelets (cells/μL) and ANC (cells/μL)). | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biller LH, Schrag D. Diagnosis and Treatment of Metastatic Colorectal Cancer: A Review. JAMA. 2021 Feb 16;325(7):669-685. doi: 10.1001/jama.2021.0106. PMID 33591350
- [Background] Ripani P, Delp J, Bode K, Delgado ME, Dietrich L, Betzler VM, Yan N, von Scheven G, Mayer TU, Leist M, Brunner T. Thiazolides promote G1 cell cycle arrest in colorectal cancer cells by targeting the mitochondrial respiratory chain. Oncogene. 2020 Mar;39(11):2345-2357. doi: 10.1038/s41388-019-1142-6. Epub 2019 Dec 16. PMID 31844249
- [Background] Shakya A, Bhat HR, Ghosh SK. Update on Nitazoxanide: A Multifunctional Chemotherapeutic Agent. Curr Drug Discov Technol. 2018;15(3):201-213. doi: 10.2174/1570163814666170727130003. PMID 28748751